CLINICAL TRIAL: NCT00550615
Title: A Phase I/II Study of Dasatinib in Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL) (BMS Protocol 180129)
Brief Title: Dasatinib in Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0244-07-FB; BMS Protocol 180129 (Other Grant/Funding Number: Bristol-Myers Squibb Company)
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkins Lymphoma; Relapsed Non Hodgkins Lymphoma; Refractory Non Hodgkins Lymphoma; Dasatinib
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dasatinib Dose Escalation (Experimental): Phase 1 employed a standard 3+3 dose-escalation design to assess safety, MTD and dose-limiting toxicity (DLT). Maximum Tolerated Dose (MTD) was defined as the next lowest dose level below where ≥ 2/3 or ≥ 3/6 patients experience dose limiting toxicities in cycle 1.
  Interventions: Drug: Dasatinib
- Dasatinib Maximum Tolerated Dose (Experimental): Once the maximum tolerated dose is determined, an additional patients will be enrolled into the Phase II portion of this trial.
  Interventions: Drug: Dasatinib Maximum Tolerated Dose

INTERVENTIONS:
Drug: Dasatinib — Dasatinib will be orally administered once daily for 28 day cycles.
  There will be three dose cohorts for the Dasatinib in the Phase I portion of this trial. A minimum of three patients will be enrolled into each of the following dose cohorts:
  Dose cohort # 1 will be 100 mg per day Dose cohort # 2 will be 150 mg per day Dose cohort # 3 will be 200 mg per day
  The MTD will be determined in the Phase I portion of this trial.
  Other Names: Spryocel
  Arms: Dasatinib Dose Escalation
Drug: Dasatinib Maximum Tolerated Dose — An additional 29 patients using the Two-Stage Simon design will be enrolled into Phase II using the MTD determined in Phase I.
  Other Names: Spryocel
  Arms: Dasatinib Maximum Tolerated Dose

SUMMARY:
Primary Objective:

* To determine the maximum tolerated dose (MTD) of Dasatinib in relapsed or refractory non-hodgkin's lymphoma (NHL) patients and to determine the safety of Dasatinib in NHL.

Secondary Objectives:

* To assess the complete and overall response rates for all Phase I and Phase II patients and to determine overall survival and event free survival for all Phase I and Phase II patients.
* To assay the levels of kinase activity in NHL specimens and correlate this activity to patient outcomes.

DETAILED DESCRIPTION:
Primary:

* To determine the Maximum Tolerated Dose (MTD) of Dasatinib in relapsed or refractory Non-Hodgkin's lymphoma (NHL) patients and to determine the safety of Dasatinib in NHL

Secondary Objective:

* To assess the complete and overall response rates for all Phase I and Phase II patients and to assay the levels of kinase activity in NHL specimens and correlate this activity to patient outcomes.
* To determine overall survival and event free survival for all Phase I and Phase II patients.

Treatment Plan

This study has two phases of treatment, Phase I and Phase II. The Phase I portion of the trial will consist of a dose escalation plan with 3-6 patients being enrolled into each dose cohort. The doses of Dasatinib used in Phase I are 100 mg, 150 mg, and 200 mg. The dose that is found to be tolerated the best and also has the best treatment results will be used for Phase II. An additional 29 patients will be enrolled into Phase II.

All patients will receive Dasatinib in this study. Dasatinib will be administered orally (by mouth) once daily for 28 day cycles. A cycle will be considered 28 days. Dosing will be continuous with no interruptions, unless instructed to interrupt treatment by the treating physician.

The patient will be restaged after every 2 cycles of therapy, every even cycle. Therapy may continue as long as there are no clinical signs of NHL progressing and the patient is tolerating the treatment with no side effects related to the therapy. If the patient is removed from study for any reason, he/she will be followed for survival until death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-hodgkin's lymphoma that is recurrent or refractory after at least one prior therapy and for which no other potentially curative therapy is available.
* Subject, age > or = 19 years
* Performance status (ECOG) 0-2
* Patients must have relapsed or refractory disease after at least one prior systemic therapy, with at least a 3 week interval from the completion of the most recent chemotherapy or radiotherapy regimen. Recover to ≤ grade 1 from all toxicities related to the prior treatments is required.
* Patients must be ineligible or relapsed after an autologous or allogeneic stem cell transplant if clinically appropriate.
* Adequate Laboratory Parameters:

  * ANC ≥ 1000/μL
  * Platelet count ≥ 50,000/μL
  * Total bilirubin < 2.0 times the institutional upper limit of normal (ULN)
  * Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN
  * Serum creatinine < 2.0 times the institutional ULN
  * PTT within institutional normal limits
* Ability to take oral medication (dasatinib must be swallowed whole)
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (sensitivity < or = 25IU HCG/L) within 72 hours prior to the start of study drug administration
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 6 months after study drug is stopped
* Signed written informed consent including HIPAA according to institutional guidelines

Exclusion Criteria:

* No malignancy [other than the one treated in this study] which required systemic treatment within the past 3 years.
* Concurrent medical condition which may increase the risk of toxicity, including:

  * Clinically significant pleural or pericardial effusion
  * Clinically-significant coagulation or platelet function disorder (e.g. known von Willebrand's disease)
* Cardiac Symptoms, consider the following:

  * Uncontrolled angina, congestive heart failure or MI within (6 months)
  * Diagnosed congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
  * Subjects with hypokalemia or hypomagnesemia if it cannot be corrected
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (< or = 3 months) significant gastrointestinal bleeding
* Concomitant Medications, consider the following prohibitions:

  * Drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib.) quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide,erythromycin, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
  * The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy.
  * Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy
  * Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
  * Patient may not be receiving any prohibited CYP3A4 inhibitors
* Women:

  * Are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks 6 months after cessation of study drug
  * Have a positive pregnancy test at baseline
  * Are pregnant or breastfeeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-09-17 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Vose, M.D., Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Internal Medicine Section of Oncology/Hematology, Omaha, Nebraska, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] Armitage JO, Weisenburger DD. New approach to classifying non-Hodgkin's lymphomas: clinical features of the major histologic subtypes. Non-Hodgkin's Lymphoma Classification Project. J Clin Oncol. 1998 Aug;16(8):2780-95. doi: 10.1200/JCO.1998.16.8.2780. PMID 9704731
- [Background] SPRYCEL (dasatinib) Tablets Prescribing Information. Bristol-Myers Squibb Company, Princeton, NJ. June 2006
- [Background] SPRYCEL® (dasatinib) BMS-354825 Bristol-Myers Squibb Investigator Brochure, Version #5, 2006.
- [Background] SPRYCEL® (dasatinib) BMS-354825 Bristol-Myers Squibb Investigator Brochure, Version #6 in print, 2006.
- [Background] Sprangers M, Feldhahn N, Herzog S, Hansmann ML, Reppel M, Hescheler J, Jumaa H, Siebert R, Muschen M. The SRC family kinase LYN redirects B cell receptor signaling in human SLP65-deficient B cell lymphoma cells. Oncogene. 2006 Aug 17;25(36):5056-62. doi: 10.1038/sj.onc.1209510. Epub 2006 Mar 27. PMID 16568084
- [Background] Zhu DM, Tibbles HE, Vassilev AO, Uckun FM. SYK and LYN mediate B-cell receptor-independent calcium-induced apoptosis in DT-40 lymphoma B-cells. Leuk Lymphoma. 2002 Nov;43(11):2165-70. doi: 10.1080/1042819021000032935. PMID 12533043
- [Background] Mahadevan D, Spier C, Della Croce K, Miller S, George B, Riley C, Warner S, Grogan TM, Miller TP. Transcript profiling in peripheral T-cell lymphoma, not otherwise specified, and diffuse large B-cell lymphoma identifies distinct tumor profile signatures. Mol Cancer Ther. 2005 Dec;4(12):1867-79. doi: 10.1158/1535-7163.MCT-05-0146. PMID 16373702
- [Background] Thompson MA, Stumph J, Henrickson SE, Rosenwald A, Wang Q, Olson S, Brandt SJ, Roberts J, Zhang X, Shyr Y, Kinney MC. Differential gene expression in anaplastic lymphoma kinase-positive and anaplastic lymphoma kinase-negative anaplastic large cell lymphomas. Hum Pathol. 2005 May;36(5):494-504. doi: 10.1016/j.humpath.2005.03.004. PMID 15948116
- [Background] Hochhaus, A. et al. Dasatinib (SPRYCEL) 50mg or 70mg BID Versus 100mg or 140mg QD in Patients with Chronic Myeloid Leukemia in Chronic Phase (CML-CP) Resistant or Intolerant to Imatinib: Results of the CA180-034 Study. American Society of Hematology, 2006 Meeting Abstracts, Part 1, Volume 108, Issue 11, November 16, 2006.
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Cohort # 1 (100 mg Per Day); Phase I Dose Cohort # 2 (150 mg Per Day); Phase I Dose Cohort # 3 (200 mg Per Day): Dasatinib will be orally administered once daily for 28 day cycles.
- Phase II Participants: Dasatinib:
  No DLT was encountered and hence the MTD was determined to be 200 mg PO daily. This was subsequently reduced to 150 mg PO daily when a higher incidence of grade 3 pleural effusions was noted.
Period: Overall Study
Arm/Group | Phase I Dose Cohort # 1 (100 mg Per Day) | Phase I Dose Cohort # 2 (150 mg Per Day) | Phase I Dose Cohort # 3 (200 mg Per Day) | Phase II Participants
Started | 3 | 3 | 10 | 22
Completed | 3 | 3 | 6 | 12
Not Completed | 0 | 0 | 4 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 3
Not completed — Not evaluable | 0 | 0 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Phase I Participants: Dasatinib will be orally administered once daily for 28 day cycles.
  There will be three dose cohorts for the Dasatinib in the Phase I portion of this trial. A minimum of three patients will be enrolled into each of the following dose cohorts:
  Dose cohort # 1 will be 100 mg per day Dose cohort # 2 will be 150 mg per day Dose cohort # 3 will be 200 mg per day
- Phase II Participants: Dasatinib:
  The MTD will be determined in the Phase I portion of this trial. An additional 29 patients using the Two-Stage Simon design will be enrolled into Phase II using the MTD determined in Phase I.
- Total: Total of all reporting groups
Arm/Group | Phase I Participants | Phase II Participants | Total
Number analyzed (Participants) | 16 | 22 | 38
Age, Continuous [Median (Full Range); unit: years] | 59 [49 to 85] | 61 [34 to 87] | 59 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 14 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Origin: Caucasian | 16 | 19 | 35
  Ethnic Origin: Black, Not Hispanic | 0 | 1 | 1
  Ethnic Origin: Hispanic | 0 | 1 | 1
  Ethnic Origin: Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 22 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Time Frame: after 1-28 day cycle of therapy
Population: Two subjects enrolled in Phase 1 of the study were never treated and not included in the analysis.
Measure: Number; unit: milligrams PO daily
Groups:
- All Phase I Participants: All participants who enrolled and treated with a minimum of 1 cycle of Dasatinib.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 14
milligrams PO daily | 200

2. Secondary Outcome: Number of Participants With Clinical Response Rates
Description: The Objective response rate (CR+PR) and the Clinical Benefit Rate (CR+PR+SD) were calculated according to revised response criteria for malignant lymphoma (Cheson) CR - Complete response is defined as: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy.
  PR - Partial response is defined as: ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses.
  SD - Stable Disease is define as: Failing to attain the criteria needed for a PR, but not fulfilling those for progressive disease.
Time Frame: after 2-28 day cycles of therapy
Population: Of the 38 participants consented only 24 for were evaluable. See the participant flow section.
Measure: Count of Participants; unit: Participants
Groups:
- Evauable Participants From Both Phases of the Trial: Response assessment was analyzed for both phases of the trial combined.
Arm/Group | Evauable Participants From Both Phases of the Trial
Number analyzed (Participants) | 24
Participants
  Objective response rate | 7
  Clinical Benefit Rate | 17

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of enrollment until 30 days after the participant completed study treatment.
Description: All doses for Phase I participants are combined as occasionally, subjects experienced adverse events leading to dose reductions so may not complete treatment at starting dose. Additionally, final adverse event reporting is most important at the maximum tolerated dose determined and use in Phase II of study.
Groups:
- Phase I Participants; Phase II Participants: All participants that were dose were monitored for adverse events.
Arm/Group | Phase I Participants | Phase II Participants
All-Cause Mortality (participants affected / at risk) | 1/14 | 4/19
Serious Adverse Events (participants affected / at risk) | 7/14 | 9/19
Other Adverse Events (participants affected / at risk) | 14/14 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Participants (N=14) | Phase II Participants (N=19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
platelet count decreased (Investigations) | 0 (0) | 1 (2)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 3 (4)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Other, Infection not specify (Infections and infestations) | 3 (3) | 1 (1)
Other, acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other, appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
cataracts (Eye disorders) | 1 (1) | 0 (0) — bilateral
Other, cellulitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Other, failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — flash
flu like symptoms (General disorders) | 1 (1) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Participants (N=14) | Phase II Participants (N=19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 6 (7)
platelet count decreased (Investigations) | 6 (6) | 11 (17)
anemia (Blood and lymphatic system disorders) | 9 (10) | 7 (13)
Fatigue (General disorders) | 6 (7) | 8 (8)
diarrhea (Gastrointestinal disorders) | 3 (4) | 9 (9)
Nausea (Gastrointestinal disorders) | 5 (6) | 7 (7)
White blood cell decreased (Investigations) | 4 (4) | 5 (12)
Neutrophil count decreased (Investigations) | 2 (4) | 6 (12)
vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3)
fever (General disorders) | 2 (2) | 5 (5)
Anorexia (Gastrointestinal disorders) | 3 (3) | 3 (3)
headache (Nervous system disorders) | 4 (4) | 2 (2)
Other - rash (Infections and infestations) | 4 (7) | 2 (2)
pericardial effusion (Cardiac disorders) | 2 (2) | 2 (3)
weakness (General disorders) | 0 (0) | 4 (4)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
chills (General disorders) | 1 (1) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Other - edema (General disorders) | 2 (2) | 3 (4)
hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Other - neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Other - cold feeling sensation (General disorders) | 0 (0) | 2 (2)
skin infection (Infections and infestations) | 2 (5) | 0 (0) — cellulitis
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
creatinine increased (Investigations) | 2 (8) | 0 (0)
Infection (Infections and infestations) | 2 (11) | 0 (0)
insomnia (Psychiatric disorders) | 2 (3) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
edema limbs (General disorders) | 2 (2) | 0 (0) — peripheral
Lung infection (Infections and infestations) | 2 (3) | 0 (0) — pneumonia
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
sinusitis (Infections and infestations) | 1 (2) | 1 (1)
gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) — stomach ache
palpitation (Cardiac disorders) | 0 (0) | 1 (1)
allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Other - alveolar inflitrates (Immune system disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other, bloated stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
cataract (Eye disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other, decrease oxygenation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
heart failure (Cardiac disorders) | 1 (1) | 0 (0) — diastolic
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — dry
dry eyes (Eye disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Other - eye swelling (Eye disorders) | 1 (1) | 0 (0)
Other, failed skin graft (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
flushing (Vascular disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
enterocolitis infection (Infections and infestations) | 0 (0) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other, generalized aches (General disorders) | 0 (0) | 1 (1)
Other, gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other - granuloma annulare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Other - hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other - Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other - Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — increased
Other - disease pain (General disorders) | 0 (0) | 1 (1)
lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Other, inflammatory skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other, intermittent diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Knee pain
Other - leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Other - loose stools (Investigations) | 1 (1) | 0 (0)
edema limbs (General disorders) | 0 (0) | 1 (1) — lower extremity
Other - Muscle cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other - muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other - muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other, myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other - pain in feet (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other - panic attacks (Psychiatric disorders) | 1 (1) | 0 (0)
genital edima (Reproductive system and breast disorders) | 0 (0) | 1 (1) — penile
genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) — scrotal
periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other - pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — lower extremity
skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other - swollen feet (General disorders) | 1 (1) | 0 (0)
Other - tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
mucosal infection (Infections and infestations) | 1 (1) | 0 (0) — thrush
Other - thyroid nodule (Endocrine disorders) | 1 (1) | 0 (0)
Other, ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Other, dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Other - vaginal atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Other - gastroenteritis (Infections and infestations) | 1 (3) | 0 (0) — viral
Other - visual disturbances (Eye disorders) | 1 (1) | 0 (0)
weight loss (Investigations) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — worsening
hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) — worsening
Other - foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — worsening

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes